CLINICAL TRIAL: NCT06021288
Title: A Randomized Controlled Study Investigating Standard Dose Continuous Renal Replacement Therapy (CRRT) Versus Low-Dose CRRT - The "Ketzerei" Trial
Brief Title: Standard Dose Continuous Renal Replacement Therapy (CRRT) Versus Low-Dose CRRT ( KETZEREI )
Acronym: KETZEREI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Münster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AnIt23-06
Record Dates: First submitted 2023-08-15; First posted 2023-09-01 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Critical Illness; Acute Kidney Injury
Keywords: Continuous renal replacement therapy
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): CRRT will be established with a draining dose (effluent dose) of 10-15ml/kg/h in pursuit of establishing a controlled azotaemia.
  Interventions: Other: Effluent dose of CRRT
- Control Group (Active Comparator): Standard of Care:
  CRRT will be established with a draining dose (effluent dose) of 25-30ml/kg/h
  Interventions: Other: Effluent dose of CRRT

INTERVENTIONS:
Other: Effluent dose of CRRT — The effluent dose of the CRRT will be performed according to study group for 7 days or up to the end of CRRT, whatever occurs first.

SUMMARY:
Acute kidney injury (AKI) is a well-recognized complication in critically ill patients, which often leads to the necessity of mechanical kidney support (CRRT).

In current therapeutic regimes, CRRT is used to strictly prevent azotaemia. Thus recent clinical observations, as well as data from animal testing suggest a link between controlled azotaemia and faster renal recovery in AKI patients.

The aim of the study is to improve renal recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years)
* Critically ill patients with AKI + in need of CRRT
* Written informed consent

Exclusion Criteria:

* Chronic dialysis dependency
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) <30 ml/min/1.73m²
* severe liver cirrhosis (Child-pugh C)
* severe acidosis (pH < 7,20 at study enrolment)
* severe hyperkalaemia (> 6mmol/l)
* Pregnancy or breastfeeding
* persons held in an institution by legal or official order
* Dependency on the investigator or center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of days alive and free from CRRT | Between Randomization and day 28

SECONDARY OUTCOMES:
Number of Adverse Events (rooted in uraemia, i.e. throwing up, seizures, uremic coma etc.) | Between randomization and day 28
Number of days with renal replacement therapy | Between randomization and day 28
Length of Intensive Care Unit (ICU) stay | Between randomization and day 28
Length of Hospital stay | Between randomization and day 28
Mortality | Day 30 after randomization
Number of new infections since randomization | From randomization until day 30
Total amount of dialysis fluid utilized adjusted for weight | From randomization until day 30
Number of patients alive and dialysis-free at day 30 | Day 30 after randomization
Presence of Major adverse kidney events (MAKE) | Day 30 after randomization
  Composite endpoint consisting of death, renal replacement therapy, and persistent severe AKI lasting for 72 hours or more
Expense of treatment (including hospital stay/all measures taken) | From randomization until day 30 after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, Study Chair — WWU Münster
Locations (2):
- Germany (2):
  - University Hospital Münster, Münster
  - Universitätsklinikum Tübingen; Universitätsklinik für Anästhesiologie und Intensivmedizin, Tübingen

REFERENCES:
- [Derived] Strauss C, Sadjadi M, von Groote T, Booke H, Schone LM, Hegner C, Wempe C, Meersch M, Gerss J, Bernard A, Haeberle HA, Rosenberger P, Rahmel T, Unterberg M, Adamzik M, Arndt C, Wulf H, Romagnoli S, Bonizzoli M, Mandarano R, Premuzic V, Andrade L, Smolentzov I, Bagshaw SM, Chawla L, Zarbock A. Randomised controlled study investigating standard dose continuous renal replacement therapy (CRRT) versus low-dose CRRT in critically ill patients with acute kidney injury (AKI): study protocol for a prospective, randomised, controlled, international, multicentre trial (the 'Ketzerei' trial). BMJ Open. 2025 Sep 22;15(9):e105459. doi: 10.1136/bmjopen-2025-105459. PMID 40983574
- [Derived] Beaubien-Souligny W, Thompson Bastin M, Teixeira JP, Cerda J, Connor MJ Jr, Dijanic Zeidman A, Garimella PS, Juncos L, Lopez-Ruiz A, Mehta R, Reis T, Rizo-Topete L, Silver SA, Da Silva JR, Speer R, Vijayan A, Wells C, Wille K, Yessayan L, Tolwani A, Neyra JA. Proceedings of the University of Alabama at Birmingham Continuous Renal Replacement Therapy Academy (2023-2024): Managing De-Escalation of Acute Renal Replacement Therapy and Optimizing Drug Dosing during Renal Replacement Therapy Transitions. Kidney360. 2025 Oct 1;6(10):1798-1809. doi: 10.34067/KID.0000000951. Epub 2025 Aug 8. PMID 40779331